CLINICAL TRIAL: NCT02250313
Title: PASCUAL (Prostate Assay Specific Clinical Utility at Launch) Study
Acronym: PASCUAL
Status: Terminated | Type: Observational
Why Stopped: Pending final analysis for termination
Sponsor: MDx Health (Industry)
Responsible Party: Sponsor
Other Study IDs: PASCUAL
Record Dates: First submitted 2014-09-16; First posted 2014-09-26 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Archived FFPE prostate biopsy core tissue to be analyzed for this study must have been collected from a previous, histologically confirmed cancer-negative biopsy. Patients were considered at risk for prostate cancer due to elevated serum PSA levels, abnormal digital rectal exam or other risk factor.
  Only archived tissues will be used in this study: no new procedures to obtain new samples from the patient will be done.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: All patients will have the tissue from their previous negative biopsy tested with the assay. Cases are defined as those subjects who receive the ConfirmMDx assay results.
- Control: All patients will have the tissue from their previous negative biopsy tested with the assay. Controls are defined as subjects who will be blinded to the ConfirmMDx assay results.

SUMMARY:
The main hypothesis of this study is to demonstrate that the use of the ConfirmMDx for Prostate Cancer test in previously biopsied patients improves urologists' patient management by reducing unnecessary repeat biopsies, attendant procedure costs, and potential adverse events in men being considered for a repeat procedure.

DETAILED DESCRIPTION:
The results of the study will reveal the clinical utility of this test by analyzing the physicians' use of negative or positive assays compared to patients managed using SOC methods without assay findings. The repeat biopsy rate at 12 months from study entry will be used for the primary endpoint analysis. All patients will be followed for 24 months from the date of the previous negative biopsy to evaluate an extended period of observation to track repeat biopsies and cancer detection.

The primary objective of this study is to demonstrate a lower repeat biopsy rate by using the negative results of ConfirmMDx for Prostate Cancer in practice rather than current SOC. All patients will have the tissue from their previous negative biopsy tested with the assay. Only data from Cases (informed of ConfirmMDx assay results) and Controls (blinded of the ConfirmMDx assay result) patients with negative test results will be used for the primary objective.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 40 to 75 years old* that underwent a previous cancer-negative prostate biopsy within 15 months and being considered for a repeat biopsy due to persistent or elevated cancer-risk factors
* The previous negative prostate biopsy must have collected a minimum of 8 tissue cores and remaining FFPE tissue from all cores should be available for testing
* Minimum tissue volume criteria of 20 microns of prostate biopsy core tissue should be available (40 microns preferable)
* The presence of HGPIN (high-grade prostatic intraepithelial neoplasia), PIA (proliferative inflammatory atrophy), or glandular inflammation reported in the first biopsy histopathology report is acceptable for entry.

Exclusion Criteria:

* Prior diagnosis of prostate cancer or cellular atypia suspicious for cancer (ASAP) in a previous biopsy histology report.
* Patients being managed by Active Surveillance for low stage prostate cancer
* Men greater than 75 years old (generally not considered for repeat biopsy)
* Most recent biopsy was a saturation biopsy (> 24 tissue cores).
* Tissue extracted using transurethral resection of the prostate (TURP) procedures rather than standard patterned biopsy core extraction.
* Subjects who had been previously tested with ConfirmMDx.

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males aged 40 to 75 years old* that underwent a previous cancer-negative prostate biopsy within 15 months and being considered for a repeat biopsy due to persistent or elevated cancer-risk factors
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate the clinical utility of the ConfirmMDx test | 2 years
  The primary objective is to demonstrate a lower repeat biopsy rate by using the negative results of ConfirmMDx for Prostate Cancer in practice rather than current SOC.

SECONDARY OUTCOMES:
Compare rebiopsy rates assay negative results in cases and controls | 2 years
  Comparison of rebiopsy rates of Cases and Controls with assay negative results at the end of follow up of 24 months from the date of the previous biopsy.
Compare rebiopsy rates in assay positive group vs standard of care | 2 years
  Comparison of rebiopsy rates in assay positive results group vs. SOC (blinded) positive assay group.
Compare rebiopsy rates of case and controls | 2 years
  Comparison of overall rates of rebiopsies of the entire Case vs. Control Cohorts
Analyse cancer detection rates | 2 years
  Analysis of cancer detection rates in ConfirmMDx positive and negative arms versus those of Controls
Evaluate clinical utility and cost savings by using the ConfirmMDx test | 2 years
  Evaluate clinical resource utilization, medical complications, and cost impact across groups
Compare rebiopsy rates assay positive results in cases and controls | 2 years
  Evaluate prostate cancer detection rates after repeat biopsy in the Case and Controls positive and negative groups at the end of 24 months after the previous negative biopsy date.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Urology Centers of Alabama, Homewood, Alabama
  - Genesis Research LLC, San Diego, California
  - Skyline Urology, Torrance, California
  - Urology Center of Colorado, Denver, Colorado
  - First Urology, PSC, Jeffersonville, Indiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Towson, Maryland
  - Michigan Institute of Urology, Troy, Michigan
  - Associated Medical Professionals of NY, Syracuse, New York
  - Oregon Urology Institute, Springfield, Oregon
  - Lancaster Urology, Lancaster, Pennsylvania
  - Carolina Urological Research Center, Myrtle Beach, South Carolina
  - Urology Associates, P.C., Nashville, Tennessee
  - Urology Clinics of North Texas, PLLC, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas